CLINICAL TRIAL: NCT03115996
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose and Multiple Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenously and Subcutaneously Administered Human Monoclonal Antibody REGN3918 in Healthy Volunteers.
Brief Title: Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of REGN3918 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R3918-HV-1659; 2016-004208-70 (EudraCT Number)
Record Dates: First submitted 2017-04-05; First posted 2017-04-14 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- REGN3918 (Cohorts 1-4 & 6a) (Experimental): Cohorts 1-4 and 6a will receive sequential ascending doses of REGN3918
  Interventions: Drug: REGN3918
- Placebo (Cohorts 1-4 & 6a) (Experimental): Cohorts 1-4 and 6a will receive placebo
  Interventions: Drug: Placebo
- REGN3918 (Cohort 5 & 6b) (Experimental): Cohort 5 and 6b will receive multiple doses of REGN3918
  Interventions: Drug: REGN3918
- Placebo (Cohort 5 & 6b) (Experimental): Cohort 5 and 6b will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN3918 — Intravenous (IV) or Subcutaneous (SC)
  Arms: REGN3918 (Cohort 5 & 6b); REGN3918 (Cohorts 1-4 & 6a)
Drug: Placebo — Matching Placebo
  Arms: Placebo (Cohort 5 & 6b); Placebo (Cohorts 1-4 & 6a)

SUMMARY:
To evaluate the safety and tolerability of single ascending intravenous (IV) and subcutaneous (SC) doses and a multiple dose regimen.

DETAILED DESCRIPTION:
Participants will be randomized to single IV or SC or multiple dose treatment with REGN3918 or matched placebo.

ELIGIBILITY:
Key Inclusion Criteria:

A subject must meet the follow criteria to be eligible for inclusion in the study:

1. Males and females from 18 to 50 years of age.
2. Subject is judged to be in good health based on medical history, physical examination, vital sign measurements and laboratory safety tests performed at screening and/or prior to administration of initial dose of study drug
3. The subject has a body mass index less than 30 kg/m2
4. Willingness to undergo vaccination and antibiotic prophylaxis against N. meningitides.

Key Exclusion Criteria:

A subject who meets any of the following criteria will be excluded from the study:

1. Any clinically significant physical examination abnormalities observed during the screening visit.
2. Hospitalization for any reason within 30 days of the screening visit
3. Persistent chronic or active recurring infection requiring treatment with antibiotics, antivirals, or antifungals.
4. Subject has a history of meningococcal infection.
5. Carriers of Neisseria meningitides based on cultures from naso-pharyngeal swabs during screening.
6. Subject has had a splenectomy.
7. Known allergy to penicillin class antibiotics
8. Known or suspected complement deficiency, or abnormal complement C3, C4 or CH50 during screening.
9. Recent (within the previous 2 months) bacterial, protozoal, viral or parasite infection requiring systemic treatment.
10. History of tuberculosis or systemic fungal diseases
11. HIV infection or HIV seropositivity at the screening visit
12. Positive HBsAg, HBcAb, or hepatitis C antibody at the screening visit
13. History of malignancy (except non-melanoma skin cancer or cervical in-situ)
14. Pregnant or breastfeeding women
15. Women of childbearing potential and men who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 6 months after the last dose

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | Up to 20 weeks
Severity of TEAEs | Up to 20 weeks

SECONDARY OUTCOMES:
Pharmacokinetic profile of REGN3918; single dose IV and SC | Up to 20 weeks
  Assessed via serum concentrations of REGN3918 over time; Area under the Curve (AUC)
Pharmacokinetic profile of REGN3918; single dose IV and repeated SC doses | Up to 20 weeks
  Assessed via serum concentrations of REGN3918 over time; peak concentration Cmax
Pharmacodynamics profile of REGN3918 | Up to 20 weeks
  Assessed by CH50 assay over time
Pharmacokinetic exploratory analysis | Up to 20 weeks
  Peak concentration Cmax
Immunogenicity of REGN3918 | Up to 20 weeks
  Assessed by measurement of anti-drug antibodies (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Covance Clinical Research Unit (CRU) Ltd., Leeds, United Kingdom

REFERENCES:
- [Derived] Devalaraja-Narashimha K, Ehmann PJ, Huang C, Ruan Q, Wipperman MF, Kaplan T, Liu C, Afolayan S, Glass DJ, Mellis S, Yancopoulos GD, Hamilton JD, MacDonnell S, Hamon SC, Boyapati A, Morton L. Association of complement pathways with COVID-19 severity and outcomes. Microbes Infect. 2023 May;25(4):105081. doi: 10.1016/j.micinf.2022.105081. Epub 2022 Dec 7. PMID 36494054